CLINICAL TRIAL: NCT04367025
Title: Efficacy and Safety of Perioperative Chemotherapy Plus PD-1 Antibody (Camrelizumabin) the Locally Advanced Adenocarcinoma of Stomach or Gastroesophageal Junction
Brief Title: Efficacy and Safety of Perioperative Chemotherapy Plus PD-1 Antibody in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Baoqing Jia, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-GC-II-007
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Camrelizumab; neoadjuvant; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOX (Active Comparator): SOX: Oxaliplatin+S-1 Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w; S-1:40~60mg Bid, d1~14, q3w; Neoadjuvant chemotherapy for 2-4 cycles, adjuvant chemotherapy for 2-4 cycles
  Interventions: Drug: Oxaliplatin; Drug: S1
- Camrelizumab+ SOX (Experimental): Camrelizumab:200mg,iv drip for 1h,d1,q3w SOX: Oxaliplatin+S-1 Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w; S-1:40~60mg Bid, d1~14, q3w; Neoadjuvant chemotherapy+ Camrelizumab for 2-4 cycles, adjuvant chemotherapy + Camrelizumab for 2-4 cycles.
  Interventions: Drug: Camrelizumab; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab: 200mg,iv drip for 1h,d1,q3w
  Other Names: SHR-1210
  Arms: Camrelizumab+ SOX
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w;
  Other Names: OXA
Drug: S1 — S-1:40~60mg Bid, d1~14, q3w;
  Arms: SOX

SUMMARY:
For locally advanced gastric cance, neoadjuvant chemotherapy can increase the resectability of tumor, and finally improve the long-term survival.

Combination of perioperative PD-1 antibody and chemotherapy for locally advanced gastric cancer could be a novel therapy to increase response rate and resectability and reduce recurrence rate. Camrelizumab（SHR-1210） in this study is a Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma and Hepatocellular carcinoma.

This study is a single center, open-label, randomized comparative phase II clinical trial to evaluate safety and efficacy of Camrelizumab in combination with perioperative chemotherapy in locally advanced adenocarcinoma of stomach or gastroesophageal junction. Differences in T cell expression were detected by single cell RNA sequencing to screen people who were more sensitive to immunotherapy.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignancies in China with incidence and mortality both ranking the 2nd among malignancies in China. Surgery is the only possible way to cure gastric cancer, however, over 80-90% of gastric cancer patients in China are in advanced stage. Locally advanced gastric cancer could be cured by multi-disciplinary therapies including surgery, chemotherapy and radiotherapy. Neoadjuvant chemotherapy can increase the resectability of tumor, and finally improve the long-term survival. However, the therapeutic effects remain unsatisfactory.

Combination of perioperative PD-1 antibody and chemotherapy for locally advanced gastric cancer could be a novel therapy to increase response rate and resectability and reduce recurrence rate. Camrelizumab in this study is a Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma and Hepatocellular carcinoma .This study is a single center, open-label, randomized comparative phase II clinical trial to evaluate safety and efficacy of Camrelizumab in combination with perioperative chemotherapy in locally advanced adenocarcinoma of stomach or gastroesophageal junction. Differences in T cell expression were detected by single cell RNA sequencing to screen people who were more sensitive to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) informed consent.
2. Age ≥ 18 years and ≤70 years.
3. ECOG Performance status 0-1.
4. Has previously untreated localized gastric or gastroesophageal junction adenocarcinoma as defined by T3 or greater primary lesion or the presence of any positive nodes - N+ (clinical nodes) without evidence of metastatic disease.
5. Patients who plan surgery after neoadjuvant chemotherapy based on clinical staging criteria.
6. Consent to send tumor tissue from biopsy or resection for PD-L1 detection and PD-L1 CPS≥1;
7. Expected survival ≥6 months;
8. Females of child bearing age must have a negative pregnancy test
9. 1）Platelet (PLT) ≥100×109/L; 2) Neutrophil count (ANC)≥1.5×l09/L; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4）WBC≥3.5×l09/L; 5) International normalized ratio (INR) ≤1.5; 5) Prothrombin time (PT) ,International Normalized Ratio（INR）and activated partial thromboplastin time (APTT) ≤1.5×ULN; 6）Total bilirubin (TBIL) level ≤1.5×ULN（patients with gilbert syndrome≤3×ULN）; 7) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN ; 10) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min;

Exclusion Criteria:

1. Patients with pathologically confirmed gastric squamous cell carcinoma, adenosquamous carcinoma, small cell carcinoma, and undifferentiated gastric cancer.
2. patients who have HER2 positive confiemed with IHC3+ or IHC2+ and FISH positive.
3. Patients with a history of t Anticancer or Experimental Therapy(Including chemotherapy, radiotherapy, hormone therapy and molecular targeted therapy)
4. The patient's cardia or pylorus is nearly obstructed, affecting eating and gastric emptying
5. Immunotherapy with previous anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies or any other antibody or drug that targets T-cell co-stimulation or immune checkpoint pathways
6. Patients have experienced or currently has other malignancies within 5 years.Except for the cured cervical carcinoma in situ,Non-melanoma skin cancer, Other tumors or cancers that have been treated radically and have shown no signs of disease for at least 5 years.
7. Peripheral neuropathy ≥ level 2（according to CTCAE 5.0）
8. Patient currently has CNS or cancerous meningitis.
9. Patients are allergic to study medication and its ingredients
10. Patients have hereditary bleeding or coagulopathy at risk of bleeding
11. Patient underwent major surgery within 4 weeks
12. Patients have taken Chinese herbal medicine or proprietary Chinese medicine for cancer treatment within two weeks
13. Patients have not recovered from complications of previous surgery.According to the CTCAE 5.0, it has not been reduced below level 1(In addition to hair loss and fatigue)
14. Patients require immunosuppressive drugs within 2 weeks or less or during the study.Exclude the following:

    A) Use of intranasal, inhaled or topical steroid(For example, intra - articular injection) B) physiological dose of steroid ( Prednisone less than 10mg per day or use equivalent dose) C) Short-term(no more than 7 day) use of steroids to prevent or treat non-autoimmune allergic diseases
15. Patients have an active or history of autoimmune disease that may recur
16. Patients have a history of interstitial lung disease or non-infectious pneumonia
17. Patients have a history of active tuberculosis
18. Patients have a history of HIV infection or other acquired, congenital immunodeficiency disease , organ transplant or stem cell transplant
19. Hepatitis B or C virus virological tests meet any of the following:

    A) HBsAg positive ,HBV-DNA≥150 copies/mL or ≥2000IU/mL B) HCV antibody positive and HCV-RNA is above the detection limit of the analysis method
20. Within 2 weeks or 2 weeks before randomization,Patients have an active or uncontrollable infection that requires systemic treatment
21. Patient vaccinated with live virus within 4 weeks
22. Patients have uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage or treatment.
23. Patients have gastrointestinal perforation or fistula within 6 months and significant clinically significant gastrointestinal bleeding before 3 months of randomization
24. Patient have intestinal obstruction, inflammatory bowel disease, extensive bowel resection, Crohn's disease, ulcerative colitis or chronic diarrhea
25. Patients have serious internal medicine diseases
26. Women who are pregnant, breast-feeding or planning to become pregnant during treatment or within 6 months after treatment ends.
27. Patients are unwilling to receive effective contraception during treatment and within 6 months after treatment ends
28. The investigator believes that the subject is not suitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | At time of surgery
  It is defined as residual tumors less than 10% after neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Objective response rate(ORR) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.
pCR | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks
  Pathological complete response
Disease-free survival (DFS) | 3years
  The time from the beginning of randomization to the recurrence of the disease or the death of the patient due to disease progression
Overall survival(OS) | From the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first,assessed up to 3 years
  The Kaplan-Meier survival from the initiation date of first cycle until death from any cause or the last follow-up date.
OSR | 3years
  overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China